CLINICAL TRIAL: NCT02495883
Title: Functional Imaging of Tremor Circuits and Mechanisms of Treatment Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Fatta B Nahab, Associate Professor of Neurosciences, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 131202; 1R01NS073683-01A1 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2015-07-13 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Essential Tremor; Tremor
Keywords: Essential Tremor; Magnetic Resonance Imaging; Therapy; Alcohol; Propranolol
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Ethanol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Essential Tremor Group (Other): Patients will be randomized to start in one of two treatment arms: 1) 50ml of 40% ethanol or 2) Propranolol SR 60-120mg. In patients who receive ethanol first, they will return for a second visit when they will receive Propranolol, and vice versa. Ethanol will be administered to participants diagnosed with Essential Tremor during the study visit, whereas patients receiving Propranolol SR will be administered daily over an estimated period of two weeks prior to the fMRI visit.
  Interventions: Other: Ethanol; Drug: Propranolol
- Health Volunteer Group (No Intervention): Healthy Volunteers will receive no interventions.

INTERVENTIONS:
Other: Ethanol — 50ml of 40% Ethanol
  Arms: Essential Tremor Group
Drug: Propranolol — Beta blocker
  Other Names: Propranolol SR; Inderal LA
  Arms: Essential Tremor Group

SUMMARY:
Essential Tremor (ET) is the most common tremor disorder, currently affecting an estimated 2.9 million Americans and leading to disability and decreased quality of life in 75% of cases. The pathophysiology of ET is poorly understood, with the source of the tremor remaining controversial since all studies show increased activity in the cerebellum (including mimicked tremor in controls), while animal models of ET using harmaline and a single human PET study implicate the inferior olivary nucleus in the brainstem.

There is evidence from the investigator's laboratory that the use of resting-state functional magnetic resonance imaging (rs-fMRI) is useful for characterizing the abnormal tremor neural network in ET compared with controls. The goal is to identify the source of the tremor, which is hypothesized to remain active during rest.

Current ET diagnostic criteria require the presence of postural and/or kinetic tremor, which are assumed to be different manifestations of the same tremor oscillator. This long-standing assumption may be incorrect based on several lines of evidence from the investigator's laboratory, and has major implications for understanding ET pathophysiology and treatment. The investigators will test the hypothesis that postural and kinetic tremors are generated through different neural mechanisms.

Treatment of ET focuses on pharmacological agents of various mechanisms and rarely deep brain stimulation of the Vim thalamus. Despite the assortment of agents used to treat ET, only ~50% of patients benefit from a particular agent. Furthermore, the mechanisms of action on tremor are not generally known. Understanding the mechanisms of action of various tremor-suppressing agents is critical for future drug development. In this proposal, the investigators plan to study the effects of ethanol (the most efficacious tremor-suppressant currently available) and propranolol (a non-specific β-adrenergic blocker with proven efficacy and unknown mechanism of action) on the tremor neural network.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ET by a Movement Disorder Neurologist.
* Tremors that improve with alcohol.
* Ability to abstain from drinking alcohol or caffeine for at least 2 days before both the screening and fMRI visits
* Over the age of 21.

Exclusion Criteria:

* Significant non-ET related abnormal findings during neurological exam.
* Presence of a tremor at rest.
* Pregnant or nursing.
* Unable to safely undergo MRI based on completion of a safety questionnaire.
* History of dementia, brain tumor, stroke, head trauma or a vascular malformation based on history or MRI findings.
* Severe active medical condition, such as cardiovascular disease, that prevents subject from lying flat for up to 120 minutes.
* Unable or unwilling to provide informed consent.
* Claustrophobia (a fear of tight spaces) or other restrictions that prevent subject from undergoing an MRI in a confined space for up to 120 minutes.
* Unable to temporarily stop taking medications that may influence liver metabolism or brain function.
* Tremors so severe that subject cannot safely and effectively undergo MRI
* Past/current problems with alcohol abuse or dependence.
* Unwillingness to take alcohol (ethanol), which is a potentially intoxicating drug
* History of deep brain stimulation or thalamotomy surgery.
* Sinus bradycardia, bronchial asthma, or a known allergy to propranolol (Inderal).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatta B Nahab, MD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Essential Tremor Group: 50ml of 40% ethanol will be administered to participants diagnosed with Essential Tremor.
  Propranolol SR 60-120mg will be administered daily to participants over an estimated period of two weeks.
  Ethanol: 50ml of 40% Ethanol
  Propranolol: Beta blocker
- Health Volunteer Group: Healthy Volunteers
Period: Overall Study
Arm/Group | Essential Tremor Group | Health Volunteer Group
Started | 32 | 24
Completed | 31 | 24
Not Completed | 1 | 0
Not completed — Excessive head motion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Essential Tremor Group | Health Volunteer Group | Total
Number analyzed (Participants) | 31 | 24 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (15.4) | 60.5 (11.5) | 62.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 17 | 8 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Total score on Montreal Cognitive Assessment (MoCA). Range of 0-30 (0-poor cognition, 30-normal cognition).
  units on a scale | 27.9 (1.7) | 28.1 (1.6) | 28.0 (1.7)
Tremor Research Group Essential Tremor Rating Scale (TETRAS) [Mean (Standard Deviation); unit: units on a scale] — Tremor Research Group Essential Tremor Rating Scale (TETRAS) is a measure of tremor severity that includes Activities of Daily Living and Performance sub scales. Total score: 112 (0-no tremor, 112-maximal tremor and disability).
  units on a scale | 37.8 (19.0) | NA (NA) — TETRAS was not done in healthy controls | 37.8 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Regions With fMRI Differences Between ET and Controls
Description: Regions that were differentially activated in ET as measured by number of statistically significant voxels (cluster size). This represents the number of activated voxels seen in the ET group that were not present in the Healthy Control group.
Time Frame: At visit 1 or 2 based on randomization table.
Population: The methodology of this trial utilizes functional MRI measures. In order to understand the significance of a group's unique brain responses, the data between the two groups (Essential Tremor vs. Healthy Controls) are statistically compared to derive regions that are unique. The output of the analyses show regions that are unique to ET.
  NOTE: Data structure cannot be provided separately for each group based on the experiment paradigm and analysis methods.
Measure: Number; unit: Number of Activated Voxels
Groups:
- All Subjects: All subject data
Arm/Group | All Subjects
Number analyzed (Participants) | 55
Number of Activated Voxels
  Right Cerebellum | 139
  Left Putamen | 93
  Right Posterior Cingulate/Thalamus | 85
  Right Sensorimotor Cortex | 74

ADVERSE EVENTS:
Time Frame: 2 study visits, each lasting up to 4 hours.
Description: Adverse events were collected in combination across both arms since the goal of the trial was to observe the differences in brain activations between the two groups (ET and healthy controls) and study the brain effects of two therapies on the ET population.
Groups:
- ET Group: Patient Cohort
- Healthy Volunteers: Control Cohort
Arm/Group | ET Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/24
Other Adverse Events (participants affected / at risk) | 0/31 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT02495883/Prot_SAP_000.pdf